CLINICAL TRIAL: NCT03818893
Title: Phase Ib/II Investigator Initiated Safety and Efficacy Clinical Trial of Combination Therapy of Intracutaneous GEN0101 With Intravenous Pembrolizmub in Patients Who Have Advanced Melanoma
Brief Title: Combination Therapy With GEN0101 and Pembrolizmub in Advanced Melanoma Patients PIb/PII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osaka University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); ISHIHARA SANGYO KAISHA,LTD. Japan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEN0101-JM005
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Advanced Melanoma
Keywords: Cancer immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New Combination Immunotherapy (Experimental): Patients will receive Pembrolizumab once every 3 weeks and a maximum of 35 doses over 105 weeks .
  The patients should be inpatient during treatment with GEN0101 in each treatment cycle and may be outpatient during off-treatment period with GEN0101, observation period, follow-up period with Pembrolizumab.
  GEN0101 in a vial will be reconstituted with 1 mL of sterile distilled water and then will be injected intracutaneously (including skin tumor site). Nonetheless, it will not be deemed as deviation if an injection has been given subcutaneously unintentionally, e.g., leakage around the peri-injection sites.
  A dose will be 60,000 mNAU in total, and 1 mL per injection site should be administered to 6 injection sites in total. For a patient, the total dose in a treatment cycle will be 360,000 mNAU (360 NAU), and the total dose over 2 treatment cycles will be 720,000 mNAU (720 NAU).
  Interventions: Drug: Combination of GEN0101 and Pembrolizmub

INTERVENTIONS:
Drug: Combination of GEN0101 and Pembrolizmub — New Combination immunotherapy GEN0101 and Pembrolizmub

SUMMARY:
This is a multi-center, open-labeled, non-randomized, single arm investigator-initiated trial to evaluate the safety and efficacy of GEN0101 and Pembrolizmub combination in patients with advanced melanoma.

DETAILED DESCRIPTION:
1. Primary Objective & Hypothesis

1. Objective: Efficacy of the combination therapy The combination therapy with intracutaneous injections of GEN0101 + intravenous infusions of Pembrolizumab is given to patients with confirmed SD or unconfirmed PD after anti-PD-1 antibody therapy. When the last subject completes Week 13 (Day 85th), the RECIST v1.1-based antitumor effect is assessed for all the subjects up to Week 17 (Day 113th) and then the ORR is calculated in both treatment groups, which are tested to examine the significant difference to historical data of KEYNOTE-002.
2. Hypothesis: The antitumor effect and the induction of antitumor immunity of the combination therapy would be enhanced.

2. Secondary Objectives & Hypothesises

1. Objectives: Efficacy and safety of the combination therapy The combination therapy with intracutaneous injections of GEN0101 + intravenous infusions of Pembrolizumab is given to patients with confirmed SD or unconfirmed PD after anti-PD-1 antibody therapy.

   When the last subject completed Week 17 (Day 113th), antitumor effect in Week 13 (Day 85th, unconfirmed) and Week 17 (Day 113th, confirmed) is assessed based on RECIST v1.1, irRC, and irRECIST for all subjects and then the ORR is calculated. Likewise, changes in individual tumor sizes in Week 13 (Day 85th, unconfirmed) and Week 17 (Day 113th, confirmed) are measured, and then percent changes in tumor sizes (percent tumor shrinkage or growth) are calculated. In each subject, the induction of antitumor immunity in Week 13 (Day 85th) is investigated with the index of activated NK cells in peripheral blood.

   When the last subject completed Week 53 (Day 365th), antitumor effect is assessed for all the subjects based on OS and RECIST v1.1, irRC, and irRECIST-based ORR, BOR and PFS, which are tested to examine significant difference to historical data of KEYNOTE-002.

   When the last subject completed Week 105 (Day 729th), antitumor effect is assessed for all the subjects based on OS and RECIST v1.1, irRC, and irRECIST-based ORR, BOR and PFS, which are tested to examine significant difference to historical data of KEYNOTE-002.

   On the basis of these results, the antitumor effect and the induction of antitumor immunity of the combination therapy is investigated. These are secondary objectives in the trial.

   As another secondary objective, AEs are investigated in all the subjects for safety evaluation of the combination therapy until the last subject completed Week 105 (Day 729th).
2. Hypothesis: The antitumor effect and the induction of antitumor immunity of the combination therapy would be enhanced and the safety would be acceptable.

3. Exploratory Objective Objective: Storage and use of samples for future exploratory evaluation

ELIGIBILITY:
Inclusion Criteria:

Patient will be eligible for this trial if all the following apply:

1. Patient has given written informed consent by themselves
2. Patient aged 20 to 85 years at the time of informed consent
3. Patient has histologically- or cytologically-confirmed melanoma
4. Patient with a diagnosis of incurable and unresectable, Stage IIIC, IIID or Stage IV advanced melanoma, showing confirmed SD or unconfirmed PD over 12-week treatment with an anti-PD-1 antibody such as nivolumab or Pembrolizumab. To be assigned a status of SD, changes in tumor measurements must be confirmed by consecutive repeat evaluations that should be performed in 4 to 6 weeks after the criteria for response are first met over 12-week of an anti-PD-1 antibody treatment.
5. Patient has a measurable tumor
6. Patient has life expectancy of at least 12 weeks after the first dose of investigational product
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening
8. Patient has met the following criteria of clinical laboratory tests at screening (1)White blood cell (WBC) count over 3,000/μL and neutrophil count over 1,500/μL (2)Platelet count over over 75,000/μL (3)Hemoglobin over 8.0 g/dL (4)AST and ALT ≤ 2.5 × upper limit of normal (ULN) (5)Total bilirubin ≤ 2 × ULN (6)Serum creatinine ≤ 2 × ULN
9. LDH is not higher than the 2-fold of the upper limit of the institutional reference.
10. A female patient of childbearing potential (a premenopausal woman, a woman with medically or drug-induced amenorrhea, and a woman with no history of sterilization), who has agreed to use appropriate contraception, e.g., the barrier method and a total abstinence, during the trial treatment until 3 months passed after completion of the trial treatment. A male patient who has agreed to use appropriate contraception, e.g., the barrier method and a total abstinence, during the above period.

Exclusion Criteria:

Patient will be excluded from participation if any of the following apply:

1. Patient has brain metastases. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging* (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
2. Patient has showed positive reaction in a prick testing for GEN0101
3. A patient who has the mutant BRAF gene in a tumor biopsy.
4. A patient who has current pneumonitis.
5. Patient concurrently has an active infection requiring systemic therapy.
6. Patient has received other systemic anticancer therapy than an anti-PD-1 antibody therapy such as nivolumab, Pembrolizumab, or local IFN-beta therapy within 3 weeks before the time of informed consent (or within 6 weeks before the time of the informed consent for a patient who received nitrosourea or mitomycin C)
7. Patient has received another unapproved drug other than anti-PD-L1 antibody within 4 weeks before the time of informed consent
8. Patient has intraocular (uveal) melanoma
9. Patient has or had another malignant tumor than melanoma. However, this criterion does not apply to a patient who has experienced neither recurrence nor metastasis for at least 5 years at the time of informed consent.
10. Patient has received systemic corticosteroid or systemic immunosuppressant within 1 week before the first dose of investigational product. However, this criterion does not apply to a patient who has been on long-term (>6-month) treatment at a low dose (equivalent to oral prednisolone under 10 mg/day) or who received prophylactic immunosuppressant against contrast media allergy.
11. Patient has received a live vaccine within 30 days before registration
12. Patient has enrolled in another clinical trial and received an investigational product within 4 months before the first dose of investigational product, or patient has intended to be enrolled in another clinical trial in parallel with this clinical trial
13. A patient who has an active TB infection.
14. Female patient is pregnant (including one with positive results from a pregnancy test at screening), lactating, or intending to become pregnant during participation in this trial and before 3 months have passed after completion of this trial. However, this criterion does not apply to a patient who will stop lactating (from the date of informed consent until 30 days passed after the last treatment). Of note, female patients should undergo a beta-HCG test to demonstrate pregnancy status. Male patient who does not agree to use appropriate contraception such as the barrier method and a total abstinence during this trial until 3 months passed after the completion of this trial. (Detailed method is described in 5.7 Contraception)
15. Patient has psychiatric disease considered to be a potential concern from the viewpoints of follow-up and protocol adherence
16. Patient had given autografting or allografting of organ or tissue (receiving an immunosuppressant)
17. Patient has over 10%-shorter prothrombin time (PT) compared to lower limit of normal (LLN) or over 1.5-fold longer activated partial thromboplastin time (APTT) compared to ULN at screening
18. Patient has showed positive reaction to any of HBs antigen, HCV antibody, HIV-1 antibody, or HIV-2 antibody at screening. However, even if it is positive for HCV antibody, it should not be excluded when HCV RNA test is negative.
19. Patient is considered ineligible for this trial by the investigator or the sub-investigators

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR), central review | until Week17 (Day113th)
  As overall tumor response in all the tumors in each subject, the ORR is calculated based on the assessment results in Week 9 (Day 57th), Week 13 (Day 85th) and Week 17 (Day 113th) as confirmatory assessment.

SECONDARY OUTCOMES:
Overall response rate (ORR) and Best overall response (BOR), investigator assessment and central review | until Week 105 (Day 729th)
  In all the tumors in each subject, the RECIST v1.1-based, the irRC-based and the irRECIST-based overall tumor response is assessed by the site investigator until Week 105 (Day 729th). Then, based on the assessment results, the ORR and BOR are calculated.
Percent change in individual tumor sizes | Until Week 105 (Day 729th)
  Until Week 105 (Day 729th) in each subject, the size of each tumor is calculated by the longest diameter the perpendicular diameter of each tumor, and then percent changes in individual tumor sizes (percent shrinkage or growth) and the local Response Rates are calculated
Progression free survival (PFS) | Until Week 105 (Day 729th)
  When the last subject completed Week 22 (Day 148th) (and Week 26 as confirmatory assessment of PD) and Week 53 (Day 365th) and Week 105 (Day 729th) of GEN0101, the RECIST v1.1-based PFS is assessed for all the subjects, where the assessment results in Week 8 should not be used and the central assessment results since Week 13 (Day 85th) only are used for all the subjects.
Overall survival (OS) | Until Week 105 (Day 729th)
  When the last subject completes Week 22 (Day 148th) and Week 53 (Day 365th) and Week 105 (Day 729th) of GEN0101, OS is calculated for all the subjects.
Induction of antitumor immunity | Week 13 (Day 85th)
  In Week 9 (Day 57th) and Week 13 (Day 85th) of GEN0101 in each subject, the induction of antitumor immunity after the combination therapy is investigated with the index of peripheral blood activated NK cells.
Adverse Events | up to Week 105 (Day 729th)
  AEs occurring in each subject up to Week 105 (Day 729th) of GEN0101 are evaluated with CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi Tanemura, Lecture, Principal Investigator — Osaka University Hospital
Locations (7):
- Japan (7):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Kumamoto University Hospital, Kuramoto, Kumamoto
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - Tokyo Medical and Dental University, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Osaka International Cancer Institute, Osaka

IPD SHARING:
Plan to Share IPD: No